CLINICAL TRIAL: NCT01155908
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of 10 mg Amlodipine Besylate/20 mg Benazepril Hydrochloride Capsules in Healthy Adult Male Volunteers Under Non-fasting (Fed) Conditions
Brief Title: Bioequivalence Study of 10 mg Amlodipine Besylate/ 20 mg Benazepril Hydrochloride Capsules of Dr.Reddys Laboratories Limited Under Non-fasting (Fed) Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Senior Manager -Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA15736
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioavailability; 10 mg Amlodipine besylate/20 mg benazepril hydrochloride capsules; Crossover
MeSH Terms: interventions — benazepril; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine Besylate/Benazepril Hydrochloride (Experimental): 10 mg Amlodipine Besylate/20 mg Benazepril Hydrochloride Capsules of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Amlodipine Besylate / Benazepril Hydrochloride
- Lotrel (Active Comparator): Lotrel® (10 mg Amlodipine Besylate / 20 mg Benazepril Hydrochloride Capsules) of Novartis
  Interventions: Drug: Amlodipine Besylate / Benazepril Hydrochloride

INTERVENTIONS:
Drug: Amlodipine Besylate / Benazepril Hydrochloride — 10 mg Amlodipine Besylate / 20 mg Benazepril Hydrochloride Capsules
  Other Names: Lotrel® (10 mg Amlodipine Besylate / 20 mg Benazepril; Hydrochloride Capsules)

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Dr. Reddy's Laboratories, Ltd. and Lotrel®) 10 mg amlodipine besylate/20 mg benazepril hydrochloride capsules, under non-fasting (fed) conditions.

DETAILED DESCRIPTION:
Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Dr. Reddy's Laboratories, Ltd. and Novartis (Lotrel®) 10 mg Amlodipine Besylate / 20 mg Benazepril Hydrochloride Capsules in Healthy Adult Male Volunteers under non-fasting (fed) Conditions

ELIGIBILITY:
Inclusion Criteria:

- Healthy adult male volunteers of 18-55 years of age;

* Weighing at least 60 kg within 15% of their ideal weights (Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company 1983)
* Medically healthy subjects with clinically normal laboratory profiles and ECGs;
* Voluntarily consent to participate in the study.

Exclusion Criteria:

- History or presence of significant cardiovascular, pulmonary, hepatic renal, hematologic,gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.

* History or presence of:

  * alcoholism or drug abuse within the past year;
  * hypersensitivity or idiosyncratic reaction to amlodipine or other calcium channel blockers;
  * hypersensitivity or idiosyncratic reaction to benazepril HCl, benazeprilat or other ACE inhibitors.
  * angioedema or anaphylactic reaction to any substance;
* Subjects whose sitting blood pressure is less than 110/60 mmHg at screening or 100/55 mmHg before dosing.
* Subjects whose pulse is lower than 55 b.p.m. at screening or 50 b.p.m. prior to dosing.
* Subjects who have used any drugs or substances known to be strong inhibitors of CYP enzymes (formerly known as cytochrome P450 enzymes) within 10 days prior to the first dose.
* Subjects who have used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
* Subjects who have vomited, who have experienced diarrhea or who have undergone vigorous and prolonged exercise (without drinking) within 24 hours prior to dosing.
* Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who, through completion of the study, would have donated in excess of: 500 mL of blood in 14 days; 1500 mL of blood in 180 days; 2500 mL of blood in 1 year.
* Subjects who have participated in another clinical trial within 28 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2005-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Bioavailability based on Cmax and AUC parameters | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, M.D, Principal Investigator — MDS Pharma Services